CLINICAL TRIAL: NCT03732599
Title: Comparison Between Standard Deep Anterior Lamellar Keratoplasty (S-DALK) and Intralase Enabled Deep Anterior Lamellar Keratoplaty (IE-DALK)
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: University of Toronto (Other)
Collaborators: Kensington Eye Institute (Other); University Health Network, Toronto (Other); Unity Health Toronto (Other); Sunnybrook Health Sciences Centre (Other); Applied Health Research Centre (Other)
Responsible Party: Principal Investigator, Neera Singal, Director of Cornea and Refractive Surgery, Kensington Eye Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 30457
Record Dates: First submitted 2018-07-10; First posted 2018-11-06 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: DALK Corneal Transplant; Keratoconus; Scar
MeSH Terms: conditions — Keratoconus; Cicatrix

STUDY DESIGN:
Intervention Model Description: This is a randomize study, in which half of the participants will be receiving either the standard deep anterior lamellar keratoplasty (DALK) (with a blade) technique or the femtosecond laser technique that creates the initial incisions instead of a blade.
Who Masked: Care Provider
Masking Description: Technologists who do the vision testing on participants are "masked" as to which "arm" the participant was randomized
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard DALK (Active Comparator): Standard (with the use of a blade) deep anterior lamellar keratoplasty (DALK), which is a partial thickness corneal transplant, which has been shown to be a safe and effective procedure.
  Interventions: Procedure: Standard Deep Anterior Keratoplasty (S-DALK)
- IE-DALK (femtosecond) (Active Comparator): Femtosecond deep anterior lamellar keratoplasty (DALK). The femotosecond laser technology allows for the creation of precise and reproducible corneal incisions.
  Interventions: Procedure: IE-DALK (femtosecond)

INTERVENTIONS:
Procedure: Standard Deep Anterior Keratoplasty (S-DALK) — Standard (with the use of a blade) deep anterior lamellar keratoplasty (DALK), which is a partial thickness corneal transplant, which has been shown to be a safe and effective procedure.
  Arms: Standard DALK
Procedure: IE-DALK (femtosecond) — Femtosecond deep anterior lamellar keratoplasty (DALK). The femotosecond laser technology allows for the creation of precise and reproducible corneal incisions.
  Arms: IE-DALK (femtosecond)

SUMMARY:
A prospective comparison between standard deep anterior lamellar keratoplasty (S-DALK) performed manually using a blade (trephine) and femtosecond laser-enabled deep anterior lamellar keratoplasty (IE DALK), where incisions are performed using the femtosecond laser.

DETAILED DESCRIPTION:
Even though corneal transplants have been around for more than 100 years, and tools to improve their surgical technique keep getting perfected, both regular and irregular postoperative astigmatism continue to be major concerns in achieving predictable visual results. Femtosecond laser technology allows for the creation of more precise incisions with more reproducible patterns, which could lead us to believe that astigmatism management and visual results should be improved with this technology. This would be the first study to prospectively analyze standard versus femtosecond laser-enabled deep anterior lamellar keratoplasties in order to elucidate their relative advantages in the quest for a gold standard.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Either advanced keratoconus or corneal scarring requiring a deep anterior lamellar keratoplasty

Exclusion Criteria:

* Previous keratoplasty
* Advanced glaucoma
* Any other retinal or optic nerve pathology that could potentially affect visual outcome
* Strabismus or amblyopia
* Significant limbal stem cell deficiency (invlolving > 3 limbal clock hours)
* Active autoimmune disease.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-04-08 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Change from preoperative topographical corneal astigmatism | preoperatively, 6, 12 and 15 months postoperatively
  Corneal astigmatism is the difference (expressed in Diopter units) of refractive power between the steep and flat corneal meridians and is measured using corneal topography. Values range between 0 and 20 diopters. Lower values represent a better outcome.

SECONDARY OUTCOMES:
Change from preoperative best-corrected distance visual acuity (BCVA) | preoperatively, 6, 12 and 15 months postoperatively.
  BCVA will be measured using an ETDRS acuity chart and recorded in logMAR (logarithm of the minimal angle of resolution) units. Value range is between -0.125 and 3 logMAR. Lower values represent a better outcome.
Change from preoperative uncorrected distance visual acuity (UCVA) | preoperatively, 6, 12 and 15 months postoperatively.
  UCVA will be measured using an ETDRS acuity chart and recorded in logMAR (logarithm of the minimal angle of resolution) units. Value range is between -0.125 and 3 logMAR. Lower values represent a better outcome.
Big-bubble success rate | 6 months postoperatively.
  This outcome represents the number of procedures where the deep anterior lamellar keratoplasty (DALK) procedure was completed using the "big bubble" surgical technique. This can either be "Yes" for successful or "No" for unsuccessful completion of this technique. Higher big-bubble success rates represent a better outcome.
Rate of conversion to penetrating keratoplasty | 6 months postoperatively.
  This outcome represents the number of failed DALK procedures (using any of the possible DALK techniques) that needed to be converted to a procedure other than DALK (a penetrating keratoplasty procedure). This can either be "Yes" for DALK failure and conversion to penetrating keratoplasty or "No" for a successful DALK procedure. Higher penetrating keratoplasty conversion rates represent a worse outcome.
Change from preoperative endothelial cell count | preoperatively, 6, 12 and 15 months postoperatively.
  This is the density of corneal endothelial cells (measured as cells per square millimeter). Value range is between 300 and 3500 cells/square millimeter. Higher values represent a better outcome.
Change from preoperative pachymetry | preoperatively, 6, 12 and 15 months postoperatively.
  This represents corneal thickness, measured in microns. Value ranges are between 200 and 800 microns. Values between 500 and 600 micron represents a good outcome.
Change from preoperative higher-order optical aberrations | preoperatively, 6, 12 and 15 months postoperatively.
  Values of total higher-order optical aberrations and coma higher-order optical aberration measured in RMS (root mean square) units. Value range is between -20 and +20 RMS. Lower absolute value represents a better outcome (values closer to zero on both the negative and positive ends).